CLINICAL TRIAL: NCT01513369
Title: Intravenous Ferric Carboxymaltose for Improvement of Metabolic Parameters and Vascular Function in T2DM-patients With Iron Deficiency
Brief Title: Ferric Carboxymaltose in Type 2 Diabetes Mellitus (T2DM) Patients With Iron Deficiency
Acronym: CLEVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLEVER-2011; 2011-005224-18 (EudraCT Number)
Record Dates: First submitted 2012-01-03; First posted 2012-01-20 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Mellitus; Iron Deficiency
Keywords: Diabetes; iron deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Iron Deficiencies; Diabetes Mellitus | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ferric carboxymaltose (Experimental): Dose: according to SmPC; Duration: 12 weeks; Frequency: at week 1 and again at week 5 (if again indicated according to principal inclusion criteria); Application: intravenous
  Interventions: Drug: ferric carboxymaltose
- NaCl (0,9%) (Placebo Comparator): Duration: 12 weeks; Frequency: at week 1 and again at week 5 (if again indicated according to principal inclusion criteria); Application: intravenous
  Interventions: Drug: NaCl (0,9%)

INTERVENTIONS:
Drug: ferric carboxymaltose — Dose:according to SmPC Duration: 12 weeks; Frequency: at week 1 and again at week 5 (if again indicated according to principal inclusion criteria); Application: intravenous
  Other Names: Ferinject (marketing authorization number: 66227.00.00)
  Arms: ferric carboxymaltose
Drug: NaCl (0,9%) — Duration: 12 weeks; Frequency: at week 1 and again at week 5 (if again indicated according to principal inclusion criteria); Application: intravenous
  Arms: NaCl (0,9%)

SUMMARY:
The purpose of this study is to investigate the correlation between HbA1c and iron status in Type 2 Diabetes mellitus patients with iron deficiency by intravenous substitution of iron.

ELIGIBILITY:
T2DM patients with diagnosis of ID defined as follows:

* serum ferritin <150 ng/mL or TSAT <25% if Hb < 14 g/dL serum ferritin <100 ng/mL or TSAT <20% if Hb ≥ 14 g/dL and ≤ 15g/dL]
* HbA1c: ≥ 6.5 to < 8.5 %
* Age > 18 years
* Written informed consent has been obtained.

Exclusion Criteria:

* Continuous subcutaneous insulin infusion (CSII)
* thalassaemia
* Hb > 15 g/dL (> 9,31 mmol/L)
* Change of HbA1c of more than ±0,3 % within the last 3 months.
* known sensitivity to ferric carboxymaltose
* history of acquired iron overload
* History of erythropoietin stimulating agent, i.v. iron therapy, and/or blood transfusion in previous 12 weeks prior to randomisation
* History of oral iron therapy at doses ≥ 100 mg/day 1 week prior to randomisation. Note: Ongoing oral use of multivitamins containing iron < 75 mg/day is permitted.
* Body weight ≤ 40 kg
* CRP > 15 mg/L
* Chronic liver disease (including known active hepatitis) and/or screening alanine transaminase (ALAT) or aspartate transaminase (ASAT) > 3 x ULN (upper limit of the normal range).
* Subjects with known hepatitis B surface antigen positivity and/or Hepatitis C virus ribonucleic acid positivity.
* Vitamin B12 and/or serum folate deficiency. If deficiency corrected subject may be rescreened for inclusion.
* Subjects with known seropositivity to human immunodeficiency virus.
* Clinical evidence of current malignancy with exception of basal cell or squamous cell carcinoma of the skin, and cervical intraepithelial neoplasia.
* Currently receiving systemic chemotherapy and/or radiotherapy.
* Renal dialysis (previous, current or planned within the next 6 months).
* Renal function GFR < 30 mL/min/ 1.73m2 (severe)
* Unstable angina pectoris as judged by the Investigator; severe valvular or left ventricular outflow obstruction disease needing intervention; atrial fibrillation/flutter with a mean ventricular response rate at rest >100 beats per minute.
* Acute myocardial infarction or acute coronary syndrome, transient ischaemic attack or stroke within the last 3 months prior to randomisation.
* Coronary-artery bypass graft, percutaneous intervention (e.g., cardiac, cerebrovascular, aortic; diagnostic catheters are allowed) or major surgery, including thoracic and cardiac surgery, within the last 3 months prior to randomisation.
* Patients with a polyneuropathy without ischemia.
* Subject of child-bearing potential who is pregnant (e.g., positive human chorionic gonadotropin test) or is breast feeding.
* Any subject not willing to use adequate contraceptive precautions during the study and for up to 5 days after the last scheduled dose of study medication.
* Participation in other interventional trials
* Female subject of child-bearing potential who is pregnant (e.g., positive human chorionic gonadotropin test) or is breast feeding.
* Failure to use highly-effective contraceptive methods
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
reduction in HBA1c-levels | 12 weeks
  reduction of HbA1c from week 1 (baseline) to week 13

SECONDARY OUTCOMES:
improvement of haematological and iron status | 12 weeks
  Hb, MCV, MCH, hypochromic cells, reticulocyte Hb content, ferritin, transferrin, transferrin saturation (TSAT), sTFR, iron, hepcidin
improvement in quality of life | 12 weeks
  potential clinical improvement and improvement in quality of life (EQ5D) of patients with ID T2DM
Improvement of metabolic status | 12 weeks
  measurement of fasting glucose, fructosamine
reliability of HbA1c-measurements | 12 weeks
  measurement of HbA1c in week 0; 5 and 13
improvement in vascular function | 12 weeks
  Improvement in vascular function on the basis of the biomarker ADMA serum level
Change in used insulin dosage during study | 12 weeks
  Change in used insulin dosage during study (via patient diary)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schindler, MD, Principal Investigator — on behalf of GWT
Locations (6):
- Germany (6):
  - Gemeinschaftspraxis Dres. Grüneberg, Mehring, Stude, Herne, North Rhine-Westphalia
  - Univesitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Herz- und Diabeteszentrum NRW Ruhr-Universität Bochum, Bad Oeynhausen
  - Studienzentrum Professor Hanefeld Abakus Büropark, Dresden
  - Medizinische Hochschule Hannover Klinisches Forschungszentrum CRC, Hanover
  - Diabetesinstitut Heidelberg, Heidelberg

REFERENCES:
- [Derived] Schindler C, Birkenfeld AL, Hanefeld M, Schatz U, Kohler C, Gruneberg M, Tschope D, Bluher M, Hasslacher C, Bornstein SR. Intravenous Ferric Carboxymaltose in Patients with Type 2 Diabetes Mellitus and Iron Deficiency: CLEVER Trial Study Design and Protocol. Diabetes Ther. 2018 Feb;9(1):37-47. doi: 10.1007/s13300-017-0330-z. Epub 2017 Nov 13. PMID 29134606